CLINICAL TRIAL: NCT02988440
Title: A Phase Ib Study of PDR001 in Combination With Sorafenib in Patients With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Study of Safety and Tolerability of PDR001 in Combination With Sorafenib and to Identify the Maximum Tolerated Dose and/or Phase 2 Dose for This Combination in Advanced Hepatocellular Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPDR001G2101; 2016-004131-20 (EudraCT Number)
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; Hepatocellular carcinoma; Hepatocellular carcinoma (HCC); PDR001; liver cancer; immunotherapy liver; malignant hepatoma; Hepatocellular cancer; advanced hepatocellular carcinoma (HCC); advanced liver cancer; liver cancer progression; sorafenib; anti-PD1; first line
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — spartalizumab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PDR001 + Sorafenib (Other): PDR001 at 400 mg given intravenously every 4 weeks and sorafenib 400 mg taken orally once or twice per day (escalating doses)
  Interventions: Drug: PDR001; Drug: Sorafenib

INTERVENTIONS:
Drug: PDR001 — PDR001 will be administered intravenously
Drug: Sorafenib — Sorafenib is formulated as a tablet.

SUMMARY:
A two part study to determine the maximum tolerated dose and/or recommended phase 2 dose of PDR001 in combination with sorafenib in patients with advanced hepatocellular carcinoma in first line. There will be a dose escalation part and a dose expansion part.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced (unresectable and/or metastatic) HCC
* Patients with advanced HCC not amenable for surgical or loco-regional treatment
* At least one measureable tumor lesion that that has not been previously locally
* Patients with current cirrhotic status of Child-Pugh class A only (5-6 points with total bilirubin < 2 mg/dL for dose-escalation) with no encephalopathy and no clinical ascites (ascites controlled by diuretics is also excluded in this study).
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patient must meet required laboratory values at the screening
* Normal electrocardiogram at screening

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
* Invasion of the main portal vein and/or tumor involvement in more than 50% of the liver (applicable only for the dose-escalation part)
* Patients with Portal-caval shunts
* Prior or concomitant systemic anti-cancer treatment for advanced disease
* Systemic chronic steroid therapy (≥ 10mg/day prednisone or equivalent) or any immunosuppressive therapy 7 days prior to planned date for first dose of study treatment. Topical, inhaled, nasal and ophthalmic steroids are allowed.
* Cardiac or cardiac repolarization abnormality
* Patients with active Hepatitis B infection (HBsAg positive) that are not receiving antiviral treatment are excluded
* Patients with positive test for hepatitis C ribonucleic acid (HCV RNA)
* Loco-regional treatment within 4 weeks prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From baseline until 30 days of last dose of study treatment
  Incidence and severity of AEs and SAEs, including changes in laboratory vital signs and ECGs
Incidendence of Dose Limiting Toxicities (DLTs) | During the first 8 weeks of treatment
  A dose-limiting toxicity (DLT) was defined as an adverse event or abnormal laboratory value assessed as unrelated to disease progression, inter-current illness, or concomitant medications that met certain criteria as defined in the protocol.
Dose interruptions | Until end of treatment, assessed for a median time of 4 months
  Tolerability measured by the number of subjects who have interruptions of study treatment
Dose reductions | Until end of treatment, assessed for a median time of 4 months
  Tolerability measured by the number of subjects who have reductions of study treatment
Dose intensity | Until end of treatment, assessed for a median time of 4 months
  Tolerability measured by the dose intensity of study treatment

SECONDARY OUTCOMES:
Overall Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as per central radiology assessment by dose level | Until end of treatment, assessed for a median time of 4 months
  Overall response rate (ORR) as per the independent central radiology assessment will be summarized descriptively by dose level. The overall response rate (ORR) is defined as the proportion of patients with best overall response of CR or PR. The best overall response is the best response recorded using the independent central radiology review based on RECIST 1.1 from start of treatment until disease progression, death, start of new therapy, withdrawal of consent or cut-off date, whichever occurs first
PDR001 trough concentration | Pre-dose at Cycle 2, 3, 4, 6 , 8, 10, 12 on Day 1. Cycle=28 days
  Concentration of PDR001 in plasma
Maximum concentration (Cmax) of sorafenib | Cycle 3 Day 1 Pre-dose, 1h, 3h and 8 h post-dose. Cycle=28 days
  The maximum (peak) observed plasma, drug concentration after single dose administration.
Time to reach maximum concentration (Tmax) of sorafenib | Cycle 3 Day 1 Pre-dose, 1h, 3h and 8 h post-dose. Cycle=28 days
  The time to reach maximum (peak) plasma drug concentration after single dose administration (time)
Area under the plasma concentration-time curve of sorafenib from time zero to 8 hours after administration (AUC0-8) | Cycle 3 Day 1 Pre-dose, 1h, 3h and 8 h post-dose. Cycle=28 days
  Area under the plasma concentration-time curve of sorafenib from time zero to time 't' where t is a defined time point after administration. t=8 hours (AUC0-8)
Area Under the Plasma Concentration-time Profile (AUCtau) of sorafenib | Cycle 3 Day 1 Pre-dose, 1h, 3h and 8 h post-dose. Cycle=28 days
  Area under the plasma concentration-time curve from time zero to the end of the dosing interval tau at steady-state

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Karmanos Cancer Institute, Detroit, Michigan, United States
- Novartis Investigative Site, Montreal, Quebec, Canada
- Novartis Investigative Site, Essen, Germany
- Novartis Investigative Site, Hong Kong, Hong Kong
- Novartis Investigative Site, Rozzano, MI, Italy
- Japan (2):
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Yokohama, Kanagawa
- Novartis Investigative Site, Pamplona, Navarre, Spain
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CPDR001G2101 from Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17724